CLINICAL TRIAL: NCT03823664
Title: Assesment of Cardiorespiratory Fitness in Prediabetic,Type 2 Diabetic and Healthy Individuals
Brief Title: Cardiorespiratory Fitness in Prediabetic,Type 2 Diabetic and Healthy Individuals
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Beyza Karadüz, Physiotherapist, Hacettepe University
Other Study IDs: GO 17/793
Record Dates: First submitted 2018-12-08; First posted 2019-01-30 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Prediabetic State; Diabetes Mellitus, Type 2; Cardiorespiratory Fitness; Inflammation; Exercise Test
Keywords: prediabetes; type 2 diabetes; cardiorespiratory fitness; pulmonary functions; functional capacity; exercise capacity
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2; Inflammation | interventions — Cardiorespiratory Fitness; Respiratory Function Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Type 2 Diabetic: Fasting Plasma Glucose ≥126 mg/dL (7.0 mmol/L). OR * A1C ≥6.5% (48 mmol/mol). OR * Patients with classic symptoms of hyperglycemia or hyperglycemic crisis, a random plasma glucose ≥200 mg/dL (11.1 mmol/L).OR* 2-h Plasma Glucose ≥200 mg/dL (11.1 mmol/L) during oral glucose tolerance test*
  * American Diabetes As. (ADA) type 2 diabetes diagnosis criteria
  Interventions: Diagnostic Test: Cardiorespiratory Fitness
- Prediabetic: Fasting Plasma Glucose 100 mg/dL (5.6 mmol/L) to 125 mg/dL (6.9 mmol/L) (Impaired Fasting Glucose)* OR A1C 5.7-6.4% (39-47 mmol/mol)* OR 2-h Plasma Glucose during 75-g Oral Glucose Tolerance Test 140 mg/dL (7.8 mmol/L) to 199 mg/dL (11.0 mmol/L) (Impaired Glucose Tolerance)*
  * ADA prediabetes criteria
  Interventions: Diagnostic Test: Cardiorespiratory Fitness
- Healthy: Healthy glucose metabolism and according to endocrinology visit no health problems related or affect cardiorespiratory fitness and other parameters examined in this study.
  Interventions: Diagnostic Test: Cardiorespiratory Fitness

INTERVENTIONS:
Diagnostic Test: Cardiorespiratory Fitness — Maximal symptom limited cardiopulmonary exercise test used assessment of cardiorespiratory fitness. For pulmonary function spirometry test and maximal respiratory pressures assessed.
  Other Names: Exercise capacity; Pulmonary function

SUMMARY:
The aim of this study to investigate and compare cardiorespiratory fitness (CRF) parameters of prediabetic, type 2 diabetic and healthy individuals. CRF assessed with cardiopulmonary exercise test (CPET) which is gold standard measure of CRF. Pulmonary functions, inflammation, disease specific parameters such as HbA1c, fasting plasma glucose etc affect CRF in prediabetic and type 2 diabetics.All parameters examine in this study.

DETAILED DESCRIPTION:
This study will be participated with Type 2 diabetic,prediabetic and healthy patients. Patients' laboratory values, pulmonary function test, respiratory muscle strength, exercise capacity, physical activity level, quality of life, cardiorespiratory fitness levels will assess and record. Pulmonary function test will be assesed with CPET system, respiratory muscle strength will be evaluated with mouth pressure. Exercise capacity will be evaluated using six minute walking test, incremental shuttle walk test. And cardiorespiratory fitness will assess CPET system. Physical activity level will be evaluated trial accelerometer and International Physical Activity Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Cooperation,
* No assistance for Ambulation,
* Body Mass Index<40
* Diagnose of prediabetes/type 2 diabetes and health

Exclusion Criteria:

* Any cardiac problems,
* Uncontrolled hypertension,
* Any neurologic disease,
* Uncontrolled diabetes,
* Any orthopedic disease impairs walking, balance
* Any respiratory disease affects cardiorespiratory fitness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetic patients -> Type 2 diabetes diagnosed population, Prediabetic -> According to ADA criteria persons in prediabetic condition Healthy
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory fitness | November 2018-August 2019
  Refers to the ability of the circulatory and respiratory systems to supply oxygen to skeletal muscles during sustained physical exercise. It will be evaluated with Cardiopulmonary Exercise Test (CPET,CPX) System

SECONDARY OUTCOMES:
Functional Exercise Capacity | December 2018-August 2019
  6 Minutes Walk Test's distance, meters
Pulmonary functions | December 2018-August 209
  Forced expiratory volume in first second (FEV1)
Respiratory Muscle Strength | December 2018-August 2019
  Mouth pressures; maximal inspiratory and expiratory pressure
Maximal Exercise Capacity | December 2018-August 2019
  İncremental Shuttle Walk Test
Physical Activity Level | December 2018-August 2019
  Accelerometer
Pulmonary functions | December 2018-August 2019
  Forced vital capacity (FVC)
Pulmonary functions | December 2018-August 2019
  Peak expiratory flow (PEF)

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Calik-Kutukcu, PhD, Study Director — Hacettepe University; Hulya Arikan, Professor, Study Chair — Hacettepe University; Cemile Bozdemir-Ozel, MsC, Study Chair — Hacettepe University; Selcuk Dagdelen, Professor, Study Chair — Hacettepe University; Beyza Nur Karaduz, PT, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided